CLINICAL TRIAL: NCT00985075
Title: A Pilot Study Evaluating the Signs and Symptoms of Seasonal Allergic Rhinitis and Conjunctivitis Following Allergen Exposure in the Allergen BioCube
Brief Title: A Pilot Study Evaluating the Signs and Symptoms of Seasonal Allergic Rhinoconjunctivitis Following Exposure in the Allergen BioCube
Status: Completed | Type: Observational
Sponsor: ORA, Inc. (Industry)
Responsible Party: H. Jerome Crampton, MD, Ophthalmic Research Associates
Other Study IDs: 08-003-14
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: Allergic rhinitis; Allergic conjunctivitis
MeSH Terms: conditions — Rhinitis, Allergic; Conjunctivitis, Allergic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to evaluate ocular and nasal signs and symptoms in patients with seasonal allergic rhinoconjunctivitis following allergen exposure in the Allergen BioCube.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age;
* if female, cannot be pregnant or nursing;
* have a history of ocular and nasal allergy and a positive skin test reaction to one of the allergens tested within the past 24 months;

Exclusion Criteria:

* have a history of mild persistent, moderate or severe asthma within the preceding 5 years according to the National Heart, Blood and Lung Institute classification;
* have a compromised lung function;
* have any ocular condition that could affect the subject's health or the study parameters;
* have any presence of active ocular or sinus infection;
* have significant nasal conditions;
* have any significant illness that could be expected to interfere with the subject's health or with the study parameters
* use specified disallowed medications (topical, topical ophthalmic, systemic and/or injectable treatments and all anti-allergy therapies) during the study or appropriate pre-study washout period;
* have used an investigational drug or device within 30 days of starting the study or be concurrently enrolled in another investigational drug or device study within 30 days of the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be 18 years of age or older with a positive history of ocular and nasal allergy and a positive skin test reaction to one of the allergens tested within the past 24 months
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Ocular Itching | At specified timepoints for up to 3 hours
Conjunctival Redness | At specified timepoints for up to 3 hours
Total Ocular Symptom Score (TOSS)of ocular itching and redness
Total Nasal Symptom Score (TNSS) of nasal symptoms

SECONDARY OUTCOMES:
Ciliary and episcleral redness | At specified timepoints for up to 3 hours
Chemosis | At specified timepoints for up to 3 hours
Lid Swelling | At specified timepoints for up to 3 hours
Tearing | At specified timepoints for up to 3 hours
Nasal Itching | At specified timepoints for up to 3 hours
Sneezing | At specified timepoints for up to 3 hours
Rhinorrhea | At specified timepoints for up to 3 hours
Nasal Congestion | At specified timepoints for up to 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gomes, MS, Study Director — ORA, Inc.; Henry J. Crampton, MD, Principal Investigator — ORA, Inc.
Locations (1):
- Ophthalmic Research Associates, Inc, Andover, Massachusetts, United States